CLINICAL TRIAL: NCT07077239
Title: MAgnetic Resonance Imaging or Computed Tomography Guided Stereotactic Body Radiotherapy With Online Adaptive Technology for Minimizing Toxicity During Salvage or AdjUvaNt Radiotherapy for ProstatE Cancer (MASAMUNE)
Brief Title: Prostate Cancer Postoperative Stereotactic Body Radiotherapy With Adaptive Technology for Minimizing Toxicity
Acronym: MASAMUNE
Status: Recruiting | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 25-0627; NCI-2025-05089 (Registry Identifier: Clinical Trials Reporting Program)
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer (CRPC)
Keywords: prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Guided Stereotactic Body Radiotherapy: Patient who has elected to receive SBRT following prostatectomy: eligibility determination based on PSA, pathology, and/or Decipher score

SUMMARY:
Single-arm, prospective registry study assessing changes in acute patient-reported urinary (GU) and gastrointestinal (GI) quality of life at the 24-month post-treatment time point following magnetic resonance imaging (MRI)-guided or computed tomography (CT)-guided stereotactic body radiotherapy (SBRT) delivered to the prostate bed +/- pelvic lymph nodes. The decision to offer an adaptive treatment will be at the clinician's discretion.

DETAILED DESCRIPTION:
This project is a single-arm, prospective study assessing changes in acute patient-reported urinary (GU) and gastrointestinal (GI) quality of life at the 24-month post-treatment time point following magnetic resonance imaging (MRI)-guided or computed tomography (CT)-guided stereotactic body radiotherapy (SBRT) delivered to the prostate bed +/- pelvic lymph nodes. There is no pre-specified target enrollment for patients undergoing standard non-adaptive SBRT. The target enrollment of patients undergoing adaptive treatment is 200 patients. The rate of accrual is expected to be in the range of 40 patients per year.

ELIGIBILITY:
Inclusion Criteria

* History of histologically confirmed, clinical localized adenocarcinoma of the prostate treated with radical prostatectomy with definitive intent.
* Presence of any ONE of the following:

  1. Adverse pathologic features at the time of prostatectomy (positive surgical margin, pathologic T-stage 3-4 disease, pathologic Gleason score 8-10 disease, OR presence of tertiary Gleason grade 5 disease)
  2. Documentation of rising prostate-specific antigen on at least two consecutive draws, with the magnitude of prostate-specific antigen exceeding 0.03 ng/mL
  3. Intermediate- or high-risk Decipher genomic classifier score
  4. Identification of prostate cancer in ≥1 lymph node at the time of prostatectomy (pN+ disease)
* CT scan and MRI of the pelvis within 120 days prior to enrollment [note: (a) if patient has medical contraindication to MRI, an exemption will be granted and enrollment can proceed; (b) for patients with PSA <1.0 ng/mL, the treatment planning CT can substitute for a diagnostic CT scan; (c) a low-field, radiation planning MRI can replace the diagnostic MRI if the patient refuses or cannot obtain a high-field MRI].
* Bone scan OR advanced nuclear imaging study within 120 days prior to enrollment for patients with PSA >1.0 ng/mL.
* Age ≥ 18.

  ~. KPS ≥ 70 and/or ECOG <2.
* Ability to understand, and willingness to sign, the written informed consent

Exclusion Criteria

* Patients with any evidence of distant metastases. Note, evidence of lymphadenopathy below the level of the renal arteries can be deemed loco regional per the discretion of the investigator.

  * Patients with neuroendocrine or small cell carcinoma of the prostate
  * Prior pelvic radiotherapy
* History of Crohn's Disease, Ulcerative Colitis, or Ataxia Telangiectasia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pN0 or pN1 prostate cancer undergoing postoperative radiotherapy targeting the prostate bed +/- pelvic lymph nodes
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2035-08-01 (Estimated); Study Completion 2036-08-01 (Estimated)

PRIMARY OUTCOMES:
Genitourinary Domain Score | 5 years
  To determine the rate of 2x MCID changes in any genitourinary domain score of the patient-reported EPIC-26 QOL tool at any point between the start of treatment and 24-months following CT-guided or MRI-guided adaptive stereotactic body radiotherapy (SBRT) to the prostate bed and/or pelvic lymph nodes.

SECONDARY OUTCOMES:
Gastrointestinal Domain Score | 5 years
  To determine the rate of 2x MCID changes in any gastrointestinal domain score of the patient-reported EPIC-26 QOL tool at any point between baseline and 24 months following CT-guided or MRI-guided adaptive stereotactic body radiotherapy (SBRT) to the prostate bed and/or pelvic lymph nodes, with a comparison to historical control data for non-adaptive post-prostatectomy SBRT regimens.
Sexual Domain Score | 5 years
  To determine the rate of 2x MCID changes in any sexual domain score of the patient-reported EPIC-26 QOL tool at any point between the start of treatment and 24-months following CT-guided or MRI-guided adaptive stereotactic body radiotherapy (SBRT) to the prostate bed and/or pelvic lymph nodes, with a comparison to historical control data for non-adaptive post-prostatectomy SBRT regimens.
Change in IPSS Score | 5 years
  To quantify changes in IPSS score at 3 month intervals within the first 12 months of treatment, then at 6 month intervals thereafter until 5 years.
Long-Term Patient Reported GU Symptoms | 5 years
  To quantify long-term patient-reported GU symptoms using the EPIC-26 instrument at 6 month intervals between 24 months and 5 years.
Long-Term Patient-Reported GI Symptoms | 5 years
  To quantify long-term patient-reported GI symptoms using the EPIC-26 instrument at 6 month intervals between 24 months and 5 years.
GU and GI Adverse Events | 5 years
  To quantify rates and severity of acute physician scored GU and GI adverse events using the Common Terminology Criteria for Adverse Events (CTCAE v. 5.0) scale.
Five-year Cumulative Incidence of GU and GI Adverse Events | 5 years
  To quantify the five-year cumulative incidence of physician scored GU and GI adverse events using the CTCAE v5.0 scale.
Progression-Free Survival | 5 years
  quantify five-year progression-free survival.
Biochemical Recurrence | 5 Years
  To quantify 5-year cumulative incidence of biochemical recurrence.
Distant Metastasis-Free Survival | 5 years
  To quantify 5-year distant metastasis-free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Valle, MD, Principal Investigator — University of California at Los Angeles
Locations (1):
- University of California at Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided